CLINICAL TRIAL: NCT04551365
Title: Effects of Lifestyle Changes and Chitosan on Gut Microbiota Modulation, Body Weight and Important Health Markers in Selected Population Groups: A Double-blind, Block-randomized, Placebo-controlled Study
Brief Title: MicroFIBERgut: Effects of Lifestyle Changes and Chitosan on Gut Microbiota and Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Collaborators: Matís ohf (Unknown); Reykjalundur Rehabilitation Center (Unknown); Primex ehf (Industry)
Responsible Party: Principal Investigator, Marta Guðjónsdóttir, Assistant professor, University of Iceland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UI-MicroFIBERgut
Record Dates: First submitted 2020-07-10; First posted 2020-09-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Lifestyle
Keywords: Gut Microbiota; Chitosan; Obesity; Body Composition; Body Weight; Health Status; Lifestyle; Defecation
MeSH Terms: conditions — Obesity; Body Weight | interventions — Rehabilitation; Chitosan

STUDY DESIGN:
Intervention Model Description: Two-block, each with 2 arms; a total of 4 arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Obese patients I (Experimental): Undergoing lifestyle changes (rehabilitation) along daily intake of chitosan supplement, 4 capsules twice daily at main meals.
  Interventions: Behavioral: Lifestyle changes; Dietary Supplement: Chitosan
- Obese patients II (Placebo Comparator): Undergoing lifestyle changes (rehabilitation) along daily intake of placebo, 4 capsules twice daily at main meals.
  Interventions: Behavioral: Lifestyle changes; Other: Placebo
- Control I (Experimental): Daily intake of chitosan supplement, 4 capsules twice daily at main meals.
  Interventions: Dietary Supplement: Chitosan
- Control II (Placebo Comparator): Daily intake of placebo 4 capsules twice daily at main meals.
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Lifestyle changes — Interdisciplinary rehabilitation programmes 5 days per week, for 4-6 weeks. The aim of the rehabilitation programme is to improve lifestyle through improved planning of activities of daily life, improved planning of food intake, increased physical activity, and weight loss. The focus is on physical and mental well-being and reinforcing participation in social activities. Patients are encouraged to carry on with their lifestyle changes after dismission from the program. Total duration 14 weeks
  Other Names: Rehabilitation
  Arms: Obese patients I; Obese patients II
Dietary Supplement: Chitosan — Daily intake of chitosan supplement. Daily dose: 4 capsules(1,5 g chitosan) twice at main meals; total 3 g Duration: 12 weeks
  Arms: Control I; Obese patients I
Other: Placebo — Daily intake of placebo (Microcrystalline cellulose (MCC), and native maize food starch (FS)) Daily dose: 4 capsules(0.75 g MCC + 0.75 g FS) twice at main meals; total 3 g Duration: 12 weeks
  Arms: Control II; Obese patients II

SUMMARY:
The purpose of this study is to compare the effects of chitosan diet supplementation to a placebo supplement on changes in gut microbiota, body weight and different health parameters among different population groups, being either obese (BMI 30-50) and undertaking major changes in lifestyle (patients) or being those not undergoing any major lifestyle changes (volunteers, BMI 18.5-35).

DETAILED DESCRIPTION:
The study will be conducted as a double-blind, block randomized, placebo-controlled intervention trial to study the effects of chitosan supplementation among two women population groups (Block 1- patients with obesity undergoing lifestyle changes; Block 2-women not undergoing major lifestyle changes) on their gut microbiota composition, body weight and composition among several other health parameters (blood pressure, blood lipids, blood sugar, insulin, hs-CRP, leptin). Furthermore, additional information will be collected: Health status, mental health, physical activity level, evaluation of stool appearance and defecation frequency by means of questionnaires; physical activity tracking, changes in body composition (muscle mass, body and visceral fat); evaluation of physical performance as well as adverse effects and remarks (diary book). The overall trial time for each subject will be 15 weeks: 1 week for baseline evaluation, 12 weeks intervention period and 2 weeks follow up.Collection of data will be done at 4 timepoints: at baseline, after 2 weeks of treatment, after 12 weeks of treatment and 2 weeks after the treatment ends (follow up).

ELIGIBILITY:
Inclusion Criteria:

Block 1

* Women, 18-80 years old with BMI >30 kg/m2, maximal supine width 65 cm.
* Living in the proximity (about 60 km radius) of Reykjavik
* Ready to stop any intake of probiotics (i.e. Bio-Kult) and weight control supplement during the trial period (3.5 months)
* Undertaking major lifestyle changes (diet and physical exercise)
* Not planning pregnancy during the treatment period (3 months)

Block 2

* Women, 18-80 years old with BMI 18.5-35 kg/m2
* Living in the proximity (about 60 km radius) of Reykjavik
* Ready to stop any intake of probiotics (i.e. Bio-Kult) and weight control supplement during the trial period (3.5 months)
* Not undertaking any major changes in lifestyle
* Not planning pregnancy during the treatment period (3 months)

Exclusion Criteria:

* Eating disorders (i.e. anorexia, bulimia)
* Inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis)
* History of poorly controlled diabetes mellitus or hypertension
* Surgical procedures (abdominal and chest) or bariatric operation in the past 6 months
* History of invasive fat reduction procedure (e.g. liposuction or abdominoplasty) within the past one year
* Drug use: a) Drugs that can cause weight loss: SGLT2 inhibitors or GLP-1 analogs or other drugs simulating incretins in the digestive system for less than 3 months b) Warfarin
* Shellfish allergy
* Pregnant or breastfeeding
* Subjects taking or having taken diet pills or weight management supplements in past 30 days
* Use of antibiotics in the last 3 months

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in the Composition of the Gut Microbiota | Change from Baseline Gut Microbiota Composition at 2 weeks
  Analysis of gut microbiota composition from stool samples
Changes in the Composition of the Gut Microbiota | Change from Baseline Gut Microbiota Composition at 12 weeks
  Analysis of gut microbiota composition from stool samples
Changes in the Composition of the Gut Microbiota | Change from Baseline Gut Microbiota Composition at 14 weeks
  Analysis of gut microbiota composition from stool samples
Changes in the Body Mass Index | Change from Baseline Body Mass Index at 2 weeks
  Body mass index calculated by dividing whole body weight by the squared height (kg/m2)
Changes in the Body Mass Index | Change from Baseline Body Mass Index at 12 weeks
  Body mass index calculated by dividing whole body weight by the squared height (kg/m2)
Changes in the Waist-to-Hip ratio | Change from Baseline Waist-to-Hip ratio at 12 weeks
  Waist circumference is measured as midpoint between the lower margin of the last palpable rib and the top of the iliac crest. Hip circumference is measured around the widest portion of the buttocks. Waist-to-hip ratio calculated by dividing waist circumference measurement by the hip circumference measurement
Changes in Total Body Fat Percentage | Change from Baseline Total Body Fat Percentage at 12 weeks
  Bioelectrical Impedance Analysis
Changes in Total Body Fat Percentage (Block 1, both arms) | Change from Baseline Total Body Fat Percentage at 12 weeks
  Dual-Energy X-Ray Absorptiometry (DXA)

SECONDARY OUTCOMES:
Changes in Abdominal Fat (Block 1, both arms) | Change from Baseline Abdominal Fat at 12 weeks
  Dual-Energy X-Ray Absorptiometry (DXA)
Changes in Lean Body Mass | Change from Baseline Lean Body Mass at 12 weeks
  Bioelectrical Impedance Analysis
Changes in Lean Body Mass (Block 1, both arms) | Change from Baseline Lean Body Mass at 12 weeks
  Dual-Energy X-Ray Absorptiometry (DXA)
Changes in Long Term Blood Glucose Concentrations | Change from Baseline Long Term Blood Glucose Concentrations at 12 weeks
  Measurement of glycated hemoglobin (B-HbAc1)
Changes in Blood Glucose Concentrations | Change from Baseline Blood Glucose Concentrations at 2 weeks
  Measurement of S-Glucose
Changes in Blood Glucose Concentrations | Change from Baseline Blood Glucose Concentrations at 12 weeks
  Measurement of S-Glucose
Changes in Blood Lipide Profile | Change from Baseline Blood Lipide Profile at 2 weeks
  Measurements of S-Cholesterol, S-High-density lipoprotein (HDL) cholesterol, S-Low-density lipoprotein (LDL) cholesterol and S-Triglycerides in blood
Changes in Blood Lipide Profile | Change from Baseline Blood Lipide Profile at 12 weeks
  Measurements of S-Cholesterol, S-High-density lipoprotein (HDL) cholesterol, S-Low-density lipoprotein (LDL) cholesterol and S-Triglycerides in blood
Changes in Inflammation Marker | Change from Baseline Inflammation Marker at 2 weeks
  Measurement of high-sensitivity C-reactive protein (hs-CRP) in blood
Changes in Inflammation Marker | Change from Baseline Inflammation Marker at 12 weeks
  Measurement of high-sensitivity C-reactive protein (hs-CRP) in blood
Changes in Six Minute Walking Distance | Change from Baseline Six Minute Walking Distance at 12 weeks
  Walking distance measured with six minute walk test in 70 meters long corridor, as a measure of exercise endurance. The longer distance walked, the better exercise endurance.
Changes in Grip Strength | Change from Baseline Grip Strength at 12 weeks
  Grip-strength measurements, three trials for each hand, mean value calculated
Changes of Satiety Feeling (Block 1, both arms) | Change from Baseline Satiety Feeling at 12 weeks
  Measurements of S-Leptin in blood

OTHER OUTCOMES:
Changes of Health Status | Change from Baseline Health Status at 12 weeks
  Measured with EQ-5D-5L questionnaire developed by the EuroQol Group. The EQ-5D-5L descriptive system comprises five dimension (5D), each describing a different aspect of current health: Mobility, Self-Care, Usual Activities, Pain/Discomfort and Anxiety/Depression. Each dimension has five response levels (5L): no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. In addition EQ visual analog scale (EQ VAS) records the respondent's overall current health on a vertical VAS, where the endpoints are labelled: "The best health you can imagine" and "The worst health you can imagine".
Changes of Depression Severity | Changes from Baseline Depression Severity at 12 weeks
  Measured with the questionnaire Depression Severity Scale (PHQ-9). It is a self-administered questionnaire with 9 items, each item can be scored from 0 (not at all) to 3 (nearly every day). Total scores can range from 0 to 27. Interpretation of Depression Severity: 0-4 None; 5-9 Mild; 10-14 Moderate; 15-19 Moderately Severe; 20-27 Severe.
Changes of General Anxiety Symptoms | Changes from Baseline General Anxiety Symptoms and at 12 weeks
  Measured with the questionnaire Generalized Anxiety Disorder Scale (GAD-7). It is a self-administered questionnaire with 7 items, each item can be scored from 0 (not at all) to 3 (nearly every day). Items are summed to create a symptom severity score ranging from 0 to 21, higher scores indicating more anxiety symptoms.
Physical Activity | 12 weeks
  Physical activity tracked with "Fitbit Charge 3" activity tracker. Each week following data will be registered: Total steps; Total minutes spent on cardiac heart rate zone; Total minutes spent in fat-burn heart rate zone; Total active minutes; Total sedentary minutes. Average value of each parameter will be used as average physical activity per week.
Changes in Physical Activity | Changes from First Half (1.- 6. weeks) average Physical Activity at Second Half (7.- 12. weeks)
  Physical activity tracked with "Fitbit Charge 3" activity tracker. Each week following data will be registered: Total steps; Total minutes spent on cardiac heart rate zone; Total minutes spent in fat-burn heart rate zone; Total active minutes; Total sedentary minutes.
Physical activity level | Baseline
  Evaluated with "Saltin-Grimby" Physical Activity Level Scale. Self-administered single-item, four level questionnaire. The single question is: How much do you move and exert yourself physically during leisure time? The question refers to the past year. The four levels range from level 1 (Physically inactive) to level 4 (Regular hard physical training for competitive sports)
Changes of Defecation | Changes from Baseline Defecation at 2 weeks
  Stool frequency questioned and consistency evaluated with Bristol Stool Form Scale. Bristol Stool Form Scale is self-administered and categorizes stools in on of seven types, ranging from type 1 (hard lumps) to type 7 (watery diarrhea).
Changes of Defecation | Changes from Baseline Defecation at 12 weeks
  Stool frequency questioned and consistency evaluated with Bristol Stool Form Scale. Bristol Stool Form Scale is self-administered and categorizes stools in on of seven types, ranging from type 1 (hard lumps) to type 7 (watery diarrhea).
Changes of Defecation | Changes from Baseline Defecation at 14 weeks
  Stool frequency questioned and consistency evaluated with Bristol Stool Form Scale. Bristol Stool Form Scale is self-administered and categorizes stools in on of seven types, ranging from type 1 (hard lumps) to type 7 (watery diarrhea).

CONTACTS AND LOCATIONS:
Overall Officials: Sigurlaug Skirnisdottir, Ph.D., Study Director — Matís ohf
Locations (1):
- Reykjalundur, Rehabilitation Center, Mosfellsbaer, Iceland

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (non-personally identifiable) will be shared that underlie results in publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Generally, data will be made available six months after the publication of each study.
Access Criteria: Data sharing request will be handled by the corresponding author of each publication.

REFERENCES:
- [Derived] Runarsdottir TR, Skirnisdottir S, Thors H, Harethardottir H, Corral-Jara KF, Klonowski AM, Halldorsson ThornI, Marteinsson VThorn, Guethjonsdottir M. The Effect of Chitosan Supplementation on the Gut Microbiota and Various Health Factors in Icelandic Females: A Placebo-Controlled, Double-Blind, Randomized Trial. Mol Nutr Food Res. 2025 Oct;69(19):e70137. doi: 10.1002/mnfr.70137. Epub 2025 Jun 8. PMID 40484808